CLINICAL TRIAL: NCT06340490
Title: A Phase I Clinical Trial of RJMty19 in Treatment of Subjects With Refractory Systemic Lupus Erythematosus
Brief Title: A Study of RJMty19 in Refractory Systemic Lupus Erythematosus (SLE)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Ruishun Biotech Co., Ltd (Industry)
Collaborators: RenJi Hospital (Other); Peking University People's Hospital (Other); Changhai Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJMty19-AID002
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: off-the-shelf cell product; CAR-DNT; Cell Therapy; Autoimmune Disease
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RJMty19 (CD19-CAR-DNT Cells) (Experimental): The trial is divided into two parts: Part A is a dose escalation trial with three dose groups (5×10^6 CAR+ cells/kg, 1×10^7 CAR+ cells/kg, 2×10^7 CAR+ cells/kg at day 0), with 9-18 patients planned to be enrolled. Part B is a dose-expansion trial in which 3~6 patients will receive RJMty19 infusions at RP2D dose levels
  Interventions: Biological: RJMty19 (CD19-CAR-DNT cells)

INTERVENTIONS:
Biological: RJMty19 (CD19-CAR-DNT cells) — Lentiviral vector-transducted double negative T cells (DNT) to express anti-CD19 CAR. Prior to cellular infusion, each patient received cyclophosphamide and fludarabine lymphodepleting chemotherapy.
  Other Names: Fludarabine; Cyclophosphamide

SUMMARY:
This study is an open-label, single-arm, dose escalation and dose expansion study to evaluate the safety, maximum tolerated dose, pharmacokinetic characteristics of allogeneic CD19-CAR-DNT cells (RJMty19) after infusion, and preliminary efficacy in systemic lupus erythematosus (SLE) subjects.

DETAILED DESCRIPTION:
The dose escalation part (Part A) plans to enroll 9-18 subjects with refractory SLE receiving RJMty19 infusion to determine the maximum tolerated dose (MTD) and/or RP2D of RJMty19. The dose expansion part (Part B) plans to enroll 3-6 subjects. The Safety Review Committee (SRC) monitors the safety information of the subjects and evaluates the safety data of each dose group. To ensure the quality of the experiment, the sponsor and inverstigators will jointly discuss and formulate the clinical research plan before the formal experiment begins.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an ICF and expect to complete the subsequent follow-up.
2. Age 18～65 years old (including cut-off value), gender is not limited.
3. Diagnosed with SLE according to the 2019 EULAR/ACR version of the revised criteria.
4. Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score ≥ 8 points; Anti-nuclear antibody titer ANA≥1:80, or positive anti-dsDNA and/or anti-Sm antibodies.
5. Presence of active organ involvement.
6. Having appropriate organ function, and the laboratory test results within 7 days before the lymphodepletion must meet the following criteria:

   1. Coagulation function:

      * Fibrinogen ≥1.0 g/L;
      * Activated partial thromboplastin time ≤ 1.5 times the upper limit of normal (ULN);
      * Prothrombin time (PT) ≤ 1.5 times ULN.
   2. Liver function:

      * Glutathione aminotransferase (AST) ≤ 3 times the upper limit of normal (ULN);
      * Glutamic aminotransferase (ALT) ≤ 3 times the upper limit of normal (ULN);
      * Total bilirubin ≤ 1.5 times ULN, unless the subject has documented Gilbert syndrome;
      * Subjects with Gilbert-Meulengracht syndrome with total bilirubin ≤ 3.0 times ULN and direct bilirubin ≤ 1.5 times ULN may be included.
   3. Renal function:

      * Serum creatinine ≤ 1.5 times ULN or a creatinine clearance ≥ 60 ml/min;
   4. Complete blood count:

      * Haemoglobin ≥ 80 g/L;
      * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L;
      * Platelet count ≥ 50 x 10^9/L;
   5. Cardiopulmonary function:

      * Left ventricular ejection fraction (LVEF) ≥ 45%;
      * Oxygen saturation ≥ 91%
7. Female patients with of childbearing potential should have a negative pregnancy test during the screening period. Any male and female patients of childbearing potential must agree to use an effective contraception method for at least six months from the time that they sign the informed consent form until the end of the cell infusion. Female subjects with non-childbearing potential (meeting at least 1 of the following criteria) is described below:

   1. Have undergone a hysterectomy or bilateral oophorectomy;
   2. Medically recognised ovarian failure;
   3. Medically recognised as post-menopausal (at least 12 consecutive months of menopause without pathological or physiological cause).
8. Use of hormones and at least two standard immunosuppressants and at least one biological agent for more than six months without meeting the LLDAS criteria; or allergy, intolerance and other drug-related side effects to the components of the biological agent make it impossible for the user to continue;
9. Life expectancy greater than 6 months;
10. Confirmed presence of CD19 positive B cells in peripheral blood by flow cytometry.

Exclusion Criteria:

1. Other malignancies within 5 years prior to screening, except adequately treated non-melanoma skin cancer (basal cell carcinoma or squamous cell carcinoma) or carcinoma in situ of the cervix;
2. Major surgery requiring hospitalization within 4 weeks prior to screening or during screening;
3. History of severe drug allergies or anaphylactic constitution;
4. Renal disease: Diagnosed with active severe lupus nephritis within 8 weeks prior to screening, requiring treatment with drugs prohibited by the study protocol for the treatment of active nephritis, hemodialysis or prednisone dose ≥ 100 mg/d, or equivalent glucocorticoids for ≥14 days; Creatinine clearance rate < 60mL/min and serum creatinine > 1.5 times ULN within 1 week before lymphodepleting chemotherapy;
5. Central nervous system diseases: those with active central nervous system diseases caused by SLE or non-SLE (including epilepsy, psychosis, organic encephalopathy syndrome, cerebrovascular accident, encephalitis, central nervous system vasculitis);
6. Cardiovascular disease: unstable angina, myocardial infarction, New York Heart Association class III or IV cardiac insufficiency, refractory hypertension (The definition of refractory hypertension is: on the basis of improving lifestyle, reasonable and tolerable use of ≥3 antihypertensive drugs (including diuretics) for more than 1 month, blood pressure still not reached the target (systolic blood pressure≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg) or taking ≥4 antihypertensive drugs to effectively control blood pressure) and a history of severe arrhythmias requiring medication;
7. Positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and peripheral blood hepatitis B virus (HBV) DNA titer test higher than the lower limit of the detection value, hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA positive, human immunodeficiency virus (HIV) antibody positive, cytomegalovirus (CMV) DNA test positive, syphilis test positive;
8. Presence of active or uncontrollable infection requiring systemic treatment (other than simple urinary tract infection or upper respiratory tract infection) and currently receiving suppressive therapy for any chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria); untreated latent tuberculosis infection;
9. There is clinical evidence showing the presence of important, unstable, or uncontrolled acute or chronic diseases not caused by SLE (i.e. cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignant tumors, or infectious diseases), which researchers believe may confound the study results or expose subjects to unnecessary risks;
10. Vaccination with live or attenuated live vaccine within 1 month before screening;
11. History of/preparing to undergo organ transplantation or hematopoietic stem cell transplantation;
12. Received CAR-T therapy or other gene-modified cell therapy prior to enrolment;
13. Have received any of the following treatments for SLE:

    1. Use of therapeutic doses of corticosteroids (defined as prednisone or equivalent> 20 mg/d) within 72 hours prior to lymphodepleting chemotherapy or RJMty19 infusion;
    2. Treatment of SLE with any other clinical investigational agent within 4 weeks prior to enrollment. However, enrollment is allowed if the study treatment period is ineffective or the disease has progressed, and at least 3 half-lives have elapsed prior to enrollment;
    3. Received belimumab within 8 weeks and anti-CD20 monoclonal antibody (e.g., rituximab) within 6 months prior to screening;
    4. Blood transfusion, packed red blood cells, and platelet transfusion within 6 weeks prior to enrollment;
    5. Plasmapheresis and plasmapheresis were treated within 3 months prior to enrollment;
14. Congenital immunoglobulin deficiency;
15. Participated in other clinical studies within the previous 3 months, except for clinical studies that have been evaluated by the investigator as not interfering with the safety and efficacy of the study drug, such as non-intervention observational studies;
16. In the judgment of the investigator and/or clinical criteria, there are contraindications to any of the study procedures or other medical conditions that may expose to unacceptable risks;
17. Presence of other autoimmune diseases that may interfere with the evaluation of efficacy (including but not limited to: rheumatoid arthritis, spondyloarthritis, dermatomyositis/polymyositis, systemic sclerosis, mixed connective tissue disease, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | Up to 28 days
  To evaluate the safety, tolerability, and determine the recommended dosage of RJMty19 for SLE subjects
Maximum Tolerated Dose (MTD) | Up to 28 days
  MTD is the highest dose for DLT in ≤1/6 subjects
Incidence of abnormalities | Up to 28 days
  Incidence of abnormalities in AE/SAE/AESI/laboratory tests/electrocardiograms/vital signs.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) indicator (Cmax) | Up to 28 days
  The peak concentration of CD19-CAR-DNT cells amplified in the peripheral blood (Cmax, detected by qPCR and Flow Cytometry).
Pharmacokinetics (PK) indicator (AUC) | Up to 90 days
  CD19-CAR-DNT cells blood concentrations will be measured at different time points to evaluate the area under the curve (AUC). (AUC, detected by qPCR and Flow Cytometry)
Pharmacokinetics (PK) indicator (CAR copy numbers) | Up to 24 months
  Changes in CAR copy numbers after injection of RJMty19
Remission rate of SLE based on DORIS criteria | at 3 months, 6 months, 12 months and 24 months
  cSLEDAI=0 and PGA < 0.5
Remission rate of SLE based on LLDAS criteria | at 3 months, 6 months, 12 months and 24 months
  SLEDAI-2K ≤ 4 points without manifestations of major organ and system involvement (renal, central nervous, cardiopulmonary, vasculitis, fever); No new disease activity compared to previous assessments (SLEDAI-2K); Physician's global assessment (PGA, 0-3) ≤1; prednisone dose (or equivalent) ≤ 7.5 mg/d; Use of stable doses of immunosuppressants and approved biologics.

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Ye, MD, PhD, Principal Investigator — RenJi Hospital; Zhanguo Li, MD, PhD, Principal Investigator — Peking University People's Hospital
Locations (4):
- China (4):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality